CLINICAL TRIAL: NCT05812586
Title: Covid-19 Vaccine Boosting in a Real World Setting: Exploratory Phase 3, Cohort Randomized, Single-blind, Multi-center Study to Evaluate the Safety and Immunogenicity of a Booster Dose of Various Covid-19 Vaccines in Fully Covid-19 Vaccine-primed Subjects Regardless of the Number of Prior Booster Dose(s) Received.
Brief Title: Assessment of Immunogenicity, Safety and Reactogenicity of a Booster Dose of Various COVID-19 Vaccine Platforms in Individuals Primed With Several Regimes.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OBU-01
Record Dates: First submitted 2023-04-06; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Exploratory phase 3, cohort randomized, single-blind, multi-center study
Who Masked: Participant
Masking Description: The participants of this study will be blinded as to the vaccine booster they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Group 1: SCB-2019/Clover (Experimental): Cohort A: complete primary immunization, no previous booster dose: SCB-2019/Clover
  Interventions: Biological: SCB-2019/Clover
- Group 2: AstraZeneca/Fiocruz (Experimental): Cohort A: complete primary immunization, no previous booster dose: AstraZeneca/Fiocruz
  Interventions: Biological: AstraZeneca/Fiocruz
- Group 3: Pfizer/Wyeth (Experimental): Cohort A: complete primary immunization, no previous booster dose: Pfizer/Wyeth
  Interventions: Biological: Pfizer/Wyeth
- Group 4: SCB-2019/Clover (Experimental): Cohort B: primary immunization plus one previous booster dose:SCB-2019/Clover
  Interventions: Biological: SCB-2019/Clover
- Group 5: AstraZeneca/Fiocruz (Experimental): Cohort B: primary immunization plus one previous booster dose: AstraZeneca/Fiocruz
  Interventions: Biological: AstraZeneca/Fiocruz
- Group 6: Pfizer/Wyeth (Experimental): Cohort B: primary immunization plus one previous booster dose: Pfizer/Wyeth
  Interventions: Biological: Pfizer/Wyeth
- Group 7: SCB-2019/Clover (Experimental): Cohort C: primary immunization plus two previous booster doses: SCB-2019/Clover
  Interventions: Biological: SCB-2019/Clover
- Group 8: AstraZeneca/Fiocruz (Experimental): Cohort C: primary immunization plus two previous booster doses: AstraZeneca/Fiocruz
  Interventions: Biological: AstraZeneca/Fiocruz
- Group 9: Pfizer/Wyeth (Experimental): Cohort C: primary immunization plus two previous booster doses: Pfizer/Wyeth
  Interventions: Biological: Pfizer/Wyeth

INTERVENTIONS:
Biological: SCB-2019/Clover — SCB-2019/Clover Vaccine
  Arms: Group 1: SCB-2019/Clover; Group 4: SCB-2019/Clover; Group 7: SCB-2019/Clover
Biological: AstraZeneca/Fiocruz — AstraZeneca/Fiocruz Vaccine
  Arms: Group 2: AstraZeneca/Fiocruz; Group 5: AstraZeneca/Fiocruz; Group 8: AstraZeneca/Fiocruz
Biological: Pfizer/Wyeth — Pfizer/Wyeth Vaccine
  Arms: Group 3: Pfizer/Wyeth; Group 6: Pfizer/Wyeth; Group 9: Pfizer/Wyeth

SUMMARY:
SARS-CoV-2 is a highly transmissible and pathogenic coronavirus that emerged in late 2019 and has caused a pandemic of acute respiratory disease, collectively known as COVID-19. Given the relatively short duration of protection after vaccination or SARS-CoV-2 infection and the evolution of immune-evading strains, it is likely that the population will have to be repeatedly boosted until a "universal" Pan-Sarbecovirus vaccine is available.

SARS-CoV-2 protein subunit vaccine candidates have shown that, despite adjuvantation, their safety/reactogenicity profile seems to be preferable over mRNA or vectored vaccines, whilst inducing non-inferior immune responses (1,2).

In this regard, serious adverse events of special interest from mRNA vaccines seem to be have been substantially underestimated/underreported. In a preliminary analysis by an International consortium, the true incidence seems to be 1,250/million excess risk in vaccinees instead of the 1-2/million reported by the Department of Health and Human Services (3,4). Additionally, in a recent study, the Clover SCB-2019 protein subunit vaccine candidate has shown higher neutralizing antibodies titers against the omicron variant, when compared to an inactivated vaccine (data not published yet). Although Brazil has various vaccine platforms authorized for emergency use or licensed, such as mRNA vaccines, vector-based vaccines, inactivated vaccines, so far Brazil has no access to adjuvanted or non-adjuvanted protein-based vaccines.

This study will involve two vaccines registered in Brazil and a protein-based adjuvanted vaccine candidate, SCB-2019/Clover. Protein-based adjuvanted vaccines have the advantage of being from a known and licensed technology that can produce high quantities of vaccine at reasonable Costs of Goods. Protein-based adjuvanted vaccines have also been shown to be highly immunogenic, both in the context of COVID-19 (2,5) and other licensed vaccines (6), with long persistence of immunity and protection.

Over 80% of the Brazilian population above the age of 18 years have received a full primary vaccination and another 7% at least one dose of vaccine. The overall booster coverage is about 48% (64% of the adults) (7). Anvisa has authorized 1st and 2nd booster doses of various vaccines in line with the MoH policy which was last updated in March 2022. It can be speculated that, like in other geographies, a third booster will be recommended soon, especially to at risk populations and in the scenario of high circulation of the Omicron BA.5 strain.

This study will explore the immunogenicity, safety and reactogenicity of a booster dose of various platforms in fully primed individuals regardless of the number of booster doses they have received prior to the enrollment in the study.

This mimics the "real world scenario" at vaccination centers where individuals with different background vaccination schemes show up for "a booster". It would facilitate logistics of immunization substantially if vaccines for boosting, independent of the immunization status, could be interchangeable with respect to safety/reactogenicity and immunogenicity. This study will enroll fully-primed individuals (2 doses of either Pfizer mRNA or Oxford/AZ/Fiocruz or Sinovac/Butantan or 1 dose of Janssen vaccine) who have received their last vaccine dose at least 4 months prior to study entry and who have received either no booster, or 1 or 2 boosters. Individuals will be stratified in cohorts by number of boosters and then randomized to receive one of 3 booster vaccines (AstraZeneca/Fiocruz, Pfizer/Wyeth, SCB-2019/Clover).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccination, laboratory tests, and other study procedures.
3. Individuals are willing and able to give an informed consent, prior to screening.
4. Individuals must have completed vaccine priming, regardless of vaccine regimen. Primary vaccination and previous booster scheme data will be annotated as patient history.
5. Interval between last dose and current study dose of a minimum of 4 months and a maximum of 24 months (to optimize candidate participation).
6. Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
7. Female participants are eligible to participate in the study if not pregnant, not breastfeeding, and at least 1 of the following criteria apply:

   * Women of non-childbearing potential;
   * Women of childbearing potential (WOCBP) must have a negative urine pregnancy test prior to study vaccination. A confirmatory serum pregnancy test may be conducted at the investigator's discretion. They must be using a highly effective licensed method of birth control during the study, until 90 days after the study vaccination.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Individuals with fever >37.5°C (axillary), or any acute illness at baseline (Day 0) or within 3 days prior to randomization. Participants meeting this criterion may be rescheduled within the relevant window. Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
2. Self-reported confirmed COVID-19 infection, through RT-PCR or lateral flow test, in the last 4 weeks.
3. Individuals who did not complete the primary vaccination scheme for any licensed COVID vaccine or plan to receive another COVID-19 vaccine (other than the study vaccines) during the study period, a drug for COVID-19 prevention or treatment (e.g., drugs, monoclonal antibodies, such as Rituximab or any other anti-CD20 monoclonal antibodies during the study period.).
4. Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis, venal or arterial thrombosis, thrombocytopenia) to any component of the study vaccines (Pfizer/Wyeth, AstraZeneca/Fiocruz, CpG 1018, aluminum, or SCB-2019 components, as outlined in the latest summary of product characteristics for Pfizer/Wyeth, AstraZeneca/Fiocruz, and the IB for SCB-2019/Clover).
5. Individuals with capillary leakage syndrome or thrombosis with thrombocytopenia syndrome

   - TTS (possibly associated with vaccination with the AstraZeneca/Fiocruz vaccine).
6. Individuals who had pericarditis or myocarditis (these pathologies may be associated with the Pfizer/Wyeth vaccine, especially in young men).
7. Individuals with known bleeding disorder that, in the opinion of the investigator, contraindicate intramuscular injection.
8. Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
9. Individuals with any progressive or severe neurologic disorder, seizure disorder, or history of Guillain-Barré syndrome.
10. Individuals who received treatment with immunosuppressive therapy in the last 90 days, including cytotoxic agents or systemic corticosteroids, or planned receipt during the study period. If a short-term course of systemic corticosteroid immunosuppressive dose has been used for the treatment of acute illness, the participant should not be included in the study until corticosteroid therapy has been discontinued for at least 15 days prior to first study vaccination.

    If the participant has used an immunosuppressive dose of a depot corticosteroid, intra-muscular or intra-articular, they must wait 60 days for inclusion in the study. Inhaled nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
11. Individuals with autoimmune diseases, except: Hashimoto's thyroiditis, vitiligo, psoriasis, lupus discord and alike; HIV-positive individuals and/or on HIV treatment.
12. Individuals who have received any other investigational product within 30 days prior to Day 0 or intend to participate in another clinical study at any time during the conduct of this study.
13. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 28 days after the last vaccination.
14. Individuals who have received treatment with Rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to Day 0 or planned during the study period.
15. Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period.
16. Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant.
17. Pregnancy.
18. Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | At baseline (day 0)
  Anti-Spike IgG antibody positivity and titers (ELISA) for SARS-CoV-2 strains (Wuhan and BA.5)
Immunogenicity | At day 28 after booster dose
  Anti-Spike IgG antibody positivity and titers (ELISA) for SARS-CoV-2 strains (Wuhan and BA.5)
Safety | Throughout the study period, an average of 3 months
  Occurrence of SAEs, AESIs and severe unsolicited AEs

SECONDARY OUTCOMES:
Immunogenicity | At days 0, 28 and 84
  VNA positivity and titers for SARS-CoV-2 strains (Wuhan, BA.5)
Immunogenicity | At day 84
  Anti-Spike IgG antibody positivity and titers (ELISA) for SARS-CoV-2 strains (Wuhan, BA.5)
Safety | Over days 0-7
  Total and severe local/systemic solicited AEs

OTHER OUTCOMES:
Documentation of confirmed SARS-CoV-2 infection | At days 28 and 84
  Occurrence of confirmed episodes of COVID-19 (by RT-PCR or lateral flow test)
Additional exploratory immunogenicity | At days 0, 28 and 84 after booster dose
  VNA and Anti-Spike IgG antibody positivity and titers (ELISA) for SARS-CoV-2 strains (Wuhan and BA.5)*

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ann C Clemens, MD, phD, Study Chair — University of Oxford
Locations (2):
- Brazil (2):
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CEPCLIN, Natal, Rio Grande do Norte
  - Centro de Referência para Imunobiológicos Especiais - CRIE - UNIFESP, São Paulo

REFERENCES:
- [Derived] Ann Costa Clemens S, Weckx L, Milan EP, Smolenov I, Clemens R. Interchangeability of different COVID-19 vaccine platforms as booster doses: A phase 3 study mimicking real-world practice. Vaccine. 2024 Jul 25;42(19):3989-3998. doi: 10.1016/j.vaccine.2024.05.009. Epub 2024 May 17. PMID 38762360